CLINICAL TRIAL: NCT02958527
Title: DRUG USE INVESTIGATION OF EFFEXOR(REGISTERED) SR CAPSULES
Brief Title: Drug Use Investigation Of Effexor (SECONDARY DATA COLLECTION STUDY; SAFETY AND EFFICACY OF EFFEXOR.UNDER JAPANESE MEDICAL PRACTICE)
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: B2411278
Record Dates: First submitted 2016-10-14; First posted 2016-11-08 (Estimated); Results first posted 2021-05-24 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2021-06

CONDITIONS: Depression/Depressed State
Keywords: Effexor; Depression; Depressed state
MeSH Terms: conditions — Depression | interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- venlafaxine: Patients with no experience of using time Effexor(venlafaxine) who will be administered time Effexor(venlafaxine)for the first
  Interventions: Drug: venlafaxine

INTERVENTIONS:
Drug: venlafaxine — The usual adult starting dosage for oral use is 37.5 mg of venlafaxine once daily, which is increased to 75 mg once daily after a meal from 1 week later. The dose may be adjusted within a range not exceeding 225 mg/day according to the patient's age and symptoms. However, the dose should be increased by 75 mg/day at intervals of not less than 1 week.
  Other Names: Effexor

SUMMARY:
SECONDARY DATA COLLECTION STUDY; SAFETY AND EFFICACY OF EFFEXOR.UNDER JAPANESE MEDICAL PRACTICE

DETAILED DESCRIPTION:
This study will be conducted under the central registration system until the number of subjects who meet the conditions for registration reaches the target number of subjects. 12 weeks from the start date. The patients who completed the 12-week treatment with this product will be observed up until Week 52.

ELIGIBILITY:
Inclusion Criteria:

* Patients with no experience of using this product who will be administered this product for the first time

Exclusion Criteria:

* Exclusion criteria are not provided in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who meet the inclusion criteria and who were registered to this study within 14 days including the start date of treatment with this product will be subjects for this study
Sampling Method: Probability Sample
Enrollment: 1408 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2020-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B2411278

RESULTS

PARTICIPANT FLOW:
Groups:
- EFFEXOR SR CAPSULES (Venlafaxine Hydrochloride): Participants who received Effexor as indicated in the approved local product document were observed for a period of 12 weeks from the start date (up until 52 weeks). The dosage can be adjusted as per physician's discretion.
Period: Overall Study
Arm/Group | EFFEXOR SR CAPSULES (Venlafaxine Hydrochloride)
Started | 1408
Completed | 1396
Not Completed | 12
Not completed — Not collected CRFs | 12

BASELINE CHARACTERISTICS:
Population: A total of 1408 participants were enrolled in this study. Of the 1396 participants who completed the study, 62 participants were excluded from the safety analysis set due to the following reasons: no adverse event information (no visit after first day of treatment)(57 participants), no drug administration (3 participants), protocol violation (2 participants).
Arm/Group | EFFEXOR SR CAPSULES (Venlafaxine Hydrochloride)
Number analyzed (Participants) | 1334
Age, Customized [Number; unit: Participants]
  <15 years | 1
  ≥15 and <65 years | 1144
  ≥65 years | 189
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 687
  Male | 647
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Drug Reactions
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to Effexor in a participant who received Effexor. A serious ADR was a ADR resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. Relatedness to Effexor was assessed by the physician.
Time Frame: 12 weeks from the start date (up until 52 weeks)
Population: The safety analysis set comprised of participants who satisfied the inclusion criteria and had received Effexor at least once.
Measure: Number; unit: Participants
Arm/Group | EFFEXOR SR CAPSULES (Venlafaxine Hydrochloride)
Number analyzed (Participants) | 1334
Participants
  ADR | 312
  Serious ADR | 4

2. Secondary Outcome: Change From Baseline in the 17-item Hamilton Rating Scale for Depression (HAM-D17) Total Scores at Pre-specified Evaluation Points
Description: HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with depression (symptoms such as depressed mood, work and activities, sleep, suicide, psychomotor agitation/retardation, appetite, sexual interest, anxiety, and somatic symptoms). The items of the HAM-D17 are rated on a scale of 0 to 2 (8 items) or from 0 to 4 (9 items), and the total score ranges from 0 to 52, higher scores indicating more severity. Change from baseline: mean score at observation minus mean score at baseline. Evaluation was performed at Week 4, 8, 12, 16, 24, 36, and 52.
Time Frame: 12 weeks from the start date ( up until 52 weeks)
Population: The efficacy analysis set comprised of participants in the safety analysis set who had effectiveness evaluation (overall evaluation by the physician based upon change in clinical symptoms and laboratory findings) at least once. Of the participants included in the efficacy analysis set (n=1312), 1259 participants had available data at baseline.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | EFFEXOR SR CAPSULES (Venlafaxine Hydrochloride)
Number analyzed (Participants) | 1259
Unit on a scale
  Week 4 (n=468): number analyzed (Participants) | 468
  Week 4 (n=468) | -6.0 (6.6)
  Week 8 (n=290): number analyzed (Participants) | 290
  Week 8 (n=290) | -9.1 (7.4)
  Week 12 (n=667): number analyzed (Participants) | 667
  Week 12 (n=667) | -12.3 (7.6)
  Week 16 (n=233): number analyzed (Participants) | 233
  Week 16 (n=233) | -11.2 (8.2)
  Week 24 (n=124): number analyzed (Participants) | 124
  Week 24 (n=124) | -12.0 (8.1)
  Week 36 (n=116): number analyzed (Participants) | 116
  Week 36 (n=116) | -12.2 (8.8)
  Week 52 (n=527): number analyzed (Participants) | 527
  Week 52 (n=527) | -15.2 (9.1)

3. Secondary Outcome: Change From Baseline in the Montgomery - Asberg Depression Rating Scale (MADRS) Total Scores at Pre-specified Evaluation Points
Description: MADRS is a clinician-administered rating scale that assesses the overall severity of depressive symptoms. The MADRS had a 10-item checklist (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts). Items are scored from 0 to 6, and the total score ranges from 0 to 60, higher scores indicating more severity. Change from baseline: mean score at observation minus mean score at baseline. Evaluation was performed at Week 4, 8, 12, 16, 24, 36, and 52.
Time Frame: 12 weeks from the start date ( up until 52 weeks)
Population: The efficacy analysis set comprised of participants in the safety analysis set who had effectiveness evaluation (overall evaluation by the physician based upon change in clinical symptoms and laboratory findings) at least once. Of the participants included in the efficacy analysis set (n=1312), 902 participants had available data at baseline.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | EFFEXOR SR CAPSULES (Venlafaxine Hydrochloride)
Number analyzed (Participants) | 902
Unit on a scale
  Week 4 (n=298): number analyzed (Participants) | 298
  Week 4 (n=298) | -7.5 (9.0)
  Week 8 (n=175): number analyzed (Participants) | 175
  Week 8 (n=175) | -11.6 (10.7)
  Week 12 (n=501): number analyzed (Participants) | 501
  Week 12 (n=501) | -15.4 (9.6)
  Week 16 (n=173): number analyzed (Participants) | 173
  Week 16 (n=173) | -15.0 (11.0)
  Week 24 (n=93): number analyzed (Participants) | 93
  Week 24 (n=93) | -13.9 (10.0)
  Week 36 (n=81): number analyzed (Participants) | 81
  Week 36 (n=81) | -15.7 (10.6)
  Week 52 (n=414): number analyzed (Participants) | 414
  Week 52 (n=414) | -19.6 (10.9)

4. Secondary Outcome: Clinical Global Impressions-Severity
Description: CGI-S is a 7-point clinician-administered rating scale that assesses overall severity of the current illness state. The score ranges from 1 to 7, higher scores indicating more affected: "1: normal, not at all ill," "2: borderline mentally ill," "3: mildly ill," "4: moderately ill," "5: markedly ill," "6: severely ill," or "7: among the most extremely ill patients." Evaluation was performed at Week 4, 8, 12, 16, 24, 36, and 52.
Time Frame: 12 weeks from the start date (up until 52 weeks)
Population: The efficacy analysis set comprised of participants in the safety analysis set who had effectiveness evaluation (overall evaluation by the physician based upon change in clinical symptoms and laboratory findings) at least once. Of the participants included in the efficacy analysis set (n=1312), a cross tabulation of the patients with available baseline CGI-S scores by CGI-S scores Week 12 and Week 52 is described.
Measure: Number; unit: Participants
Groups:
- EFFEXOR SR CAPSULES (Venlafaxine Hydrochloride) Baseline 1; EFFEXOR SR CAPSULES (Venlafaxine Hydrochloride) Baseline 2; EFFEXOR SR CAPSULES (Venlafaxine Hydrochloride) Baseline 3; EFFEXOR SR CAPSULES (Venlafaxine Hydrochloride) Baseline 4; EFFEXOR SR CAPSULES (Venlafaxine Hydrochloride) Baseline 5; EFFEXOR SR CAPSULES (Venlafaxine Hydrochloride) Baseline 6; EFFEXOR SR CAPSULES (Venlafaxine Hydrochloride) Baseline 7: Participants who received Effexor as indicated in the approved local product document were observed for a period of 12 weeks from the start date (up until 52 weeks). The dosage can be adjusted as per physician's discretion.
Arm/Group | EFFEXOR SR CAPSULES (Venlafaxine Hydrochloride) Baseline 1 | EFFEXOR SR CAPSULES (Venlafaxine Hydrochloride) Baseline 2 | EFFEXOR SR CAPSULES (Venlafaxine Hydrochloride) Baseline 3 | EFFEXOR SR CAPSULES (Venlafaxine Hydrochloride) Baseline 4 | EFFEXOR SR CAPSULES (Venlafaxine Hydrochloride) Baseline 5 | EFFEXOR SR CAPSULES (Venlafaxine Hydrochloride) Baseline 6 | EFFEXOR SR CAPSULES (Venlafaxine Hydrochloride) Baseline 7
Number analyzed (Participants) | 1 | 7 | 182 | 590 | 285 | 104 | 4
Participants
  Week 12 1: Normal, not at all ill | 0 | 2 | 19 | 56 | 9 | 7 | 1
  Week 12 2: Borderline mentally ill | 0 | 1 | 45 | 98 | 38 | 15 | 1
  Week 12 3: Mildly ill | 0 | 0 | 24 | 133 | 52 | 10 | 0
  Week 12 4: Moderately ill | 0 | 0 | 2 | 45 | 61 | 10 | 0
  Week 12 5: Markedly ill | 0 | 0 | 0 | 2 | 13 | 7 | 0
  Week 12 6: Severely ill | 0 | 0 | 0 | 0 | 1 | 5 | 0
  Week 12 7: Among the most extremely ill patients | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 52 1: Normal, not at all ill | 0 | 0 | 27 | 76 | 40 | 16 | 1
  Week 52 2: Borderline mentally ill | 0 | 2 | 33 | 92 | 47 | 14 | 0
  Week 52 3: Mildly ill | 0 | 0 | 15 | 69 | 39 | 7 | 0
  Week 52 4: Moderately ill | 0 | 0 | 0 | 21 | 14 | 2 | 0
  Week 52 5: Markedly ill | 0 | 0 | 0 | 2 | 5 | 1 | 0
  Week 52 6: Severely ill | 0 | 0 | 0 | 1 | 0 | 4 | 0
  Week 52 7: Among the most extremely ill patients | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Changes in the Clinical Global Impressions-Improvement
Description: CGI-I is a 7-point clinician-administered rating scale that assesses overall improvement of the disease/condition. The score ranges from 1 to 7, higher scores indicating more affected: was assessed as "1: markedly improved," "2: moderately improved," "3: mildly improved," "4: no change," "5: slightly worsened," "6: worsened," or "7: severely worsened." Evaluation was performed at Week 4, 8, 12, 16, 24, 36, and 52.
Time Frame: 12 weeks from the start date (up until 52 weeks)
Population: The efficacy analysis set comprised of participants in the safety analysis set who had effectiveness evaluation (overall evaluation by the physician based upon change in clinical symptoms and laboratory findings) at least once. Of the participants included in the efficacy analysis set (n=1312), those who had available data at Week 12 and 52 were evaluated.
Measure: Number; unit: Participants
Groups:
- EFFEXOR SR CAPSULES (Venlafaxine Hydrochloride) Week 12; EFFEXOR SR CAPSULES (Venlafaxine Hydrochloride) Week 52: Participants who received Effexor as indicated in the approved local product document were observed for a period of 12 weeks from the start date (up until 52 weeks). The dosage can be adjusted as per physician's discretion.
Arm/Group | EFFEXOR SR CAPSULES (Venlafaxine Hydrochloride) Week 12 | EFFEXOR SR CAPSULES (Venlafaxine Hydrochloride) Week 52
Number analyzed (Participants) | 664 | 533
Participants
  1: Markedly improved | 199 | 235
  2: Moderately improved | 175 | 178
  3: Mildly improved | 212 | 88
  4: No change | 70 | 28
  5: Slightly worsened | 5 | 3
  6: Worsened | 3 | 1
  7: Severely worsened | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks from the start date (up until 52 weeks)
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both serious and non-serious events during the study.
Arm/Group | EFFEXOR SR CAPSULES (Venlafaxine Hydrochloride)
All-Cause Mortality (participants affected / at risk) | 0/1334
Serious Adverse Events (participants affected / at risk) | 20/1334
Other Adverse Events (participants affected / at risk) | 495/1334
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EFFEXOR SR CAPSULES (Venlafaxine Hydrochloride) (N=1334)
Alcoholic pancreatitis (Gastrointestinal disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Anaphylactic shock (Immune system disorders) | 1
Pneumonia (Infections and infestations) | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Completed suicide (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Depressive symptom (Psychiatric disorders) | 1
Hypomania (Psychiatric disorders) | 1
Mania (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 2
Suicide attempt (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EFFEXOR SR CAPSULES (Venlafaxine Hydrochloride) (N=1334)
Palpitations (Cardiac disorders) | 13
Tinnitus (Ear and labyrinth disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 36
Diarrhoea (Gastrointestinal disorders) | 10
Eructation (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 3
Gastrointestinal disorder (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 76
Vomiting (Gastrointestinal disorders) | 7
Chest pain (General disorders) | 2
Feeling abnormal (General disorders) | 3
Malaise (General disorders) | 26
Thirst (General disorders) | 5
Withdrawal syndrome (General disorders) | 2
Hepatic function abnormal (Hepatobiliary disorders) | 12
Hepatic steatosis (Hepatobiliary disorders) | 2
Liver disorder (Hepatobiliary disorders) | 3
Gastroenteritis (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 2
Blood pressure increased (Investigations) | 6
Weight increased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 13
Dyslipidaemia (Metabolism and nutrition disorders) | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3
Hyperlipidaemia (Metabolism and nutrition disorders) | 4
Hyperphagia (Metabolism and nutrition disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Akathisia (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 25
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 23
Hypersomnia (Nervous system disorders) | 5
Hypoaesthesia (Nervous system disorders) | 2
Migraine (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 53
Tremor (Nervous system disorders) | 3
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 3
Anger (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 3
Hallucination, auditory (Psychiatric disorders) | 3
Hypomania (Psychiatric disorders) | 5
Initial insomnia (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 39
Intentional self-injury (Psychiatric disorders) | 3
Irritability (Psychiatric disorders) | 2
Libido decreased (Psychiatric disorders) | 2
Mania (Psychiatric disorders) | 5
Middle insomnia (Psychiatric disorders) | 6
Sleep disorder (Psychiatric disorders) | 5
Suicidal ideation (Psychiatric disorders) | 5
Dysuria (Renal and urinary disorders) | 6
Pollakiuria (Renal and urinary disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 2
Ejaculation disorder (Reproductive system and breast disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7
Night sweats (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 2
Orthostatic hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-12-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT02958527/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/27/NCT02958527/SAP_001.pdf